CLINICAL TRIAL: NCT04634071
Title: Tobacco Treatment Optimization and Preferences During Concurrent Cancer Treatment
Acronym: TTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Valentino, MD (Other)
Responsible Party: Sponsor-Investigator, Joseph Valentino, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-MULTI-34
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Cancer, Treatment-Related
Keywords: Addiction; Cancer Therapy; Tobacco; nicotine
MeSH Terms: conditions — Smoking Cessation; Neoplasms, Second Primary; Behavior, Addictive | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: This trial is a parallel design. However, it is part of a broader sequential cohort design to compare the effects of preference driven tobacco treatment upon cessation versus effects of a previous cohort from a separate randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Group 1: Varenicline, Intense Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive varenicline, counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Varenicline; Behavioral: High-intensity counseling; Drug: Nicotine Replacement Products
- Group : Varenicline, Intense Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive varenicline and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Varenicline; Behavioral: High-intensity counseling; Other: No nicotine replacement therapy
- Group 3: Varenicline, Minimal Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive varenicline, counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Varenicline; Behavioral: Low-intensity counseling; Drug: Nicotine Replacement Products
- Group 4: Varenicline, Minimal Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive varenicline and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Varenicline; Behavioral: Low-intensity counseling; Other: No nicotine replacement therapy
- Group 5: Buproprion, Intense Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive Buproprion, counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Bupropion; Behavioral: High-intensity counseling; Drug: Nicotine Replacement Products
- Group 6: Buproprion, Intense Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive Buproprion and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Bupropion; Behavioral: High-intensity counseling; Other: No nicotine replacement therapy
- Group 7: Buproprion, Minimal Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive Buproprion, counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Bupropion; Behavioral: Low-intensity counseling; Drug: Nicotine Replacement Products
- Group 8: Buproprion, Minimal Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive Buproprion and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Bupropion; Behavioral: Low-intensity counseling; Other: No nicotine replacement therapy
- Group 9: Nicotine, Intense Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive long acting nicotine replacement therapy (e.g. nicotine patch), counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Long-acting nicotine replacement therapy; Behavioral: High-intensity counseling; Drug: Nicotine Replacement Products
- Group 10: Nicotine, Intense Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive long acting nicotine replacement therapy (e.g. nicotine patch) and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Long-acting nicotine replacement therapy; Behavioral: High-intensity counseling; Other: No nicotine replacement therapy
- Group 11: Nicotine, Minimal Counselling and NRT (Experimental): Patients diagnosed with tobacco-related treatment will receive long acting nicotine replacement therapy (e.g. nicotine patch), counseling, and nicotine replacement therapy (PRN NRT). Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Long-acting nicotine replacement therapy; Behavioral: Low-intensity counseling; Drug: Nicotine Replacement Products
- Group 12: Nicotine, Minimal Counselling (Experimental): Patients diagnosed with tobacco-related treatment will receive long acting nicotine replacement therapy (e.g. nicotine patch) and counseling. Dose and frequency will be based on patient preference, smoking history and other medical factors.
  Interventions: Drug: Long-acting nicotine replacement therapy; Behavioral: Low-intensity counseling; Other: No nicotine replacement therapy

INTERVENTIONS:
Drug: Varenicline — Varenicline therapy will be 12-week course. On days 1-3 participants will receive 0.5mg once daily; days 4-7 receive 0.5mg twice daily and day 8 until the end of treatment receive 1mg twice daily.
  Other Names: Chantix
  Arms: Group 1: Varenicline, Intense Counselling and NRT; Group 3: Varenicline, Minimal Counselling and NRT; Group 4: Varenicline, Minimal Counselling; Group : Varenicline, Intense Counselling
Drug: Bupropion — Patients will begin with a dose of 150 mg every morning for 3 days. Then dosage will increase to 150 mg twice daily (morning and evening), for a total daily dose of 300 mg, for 7 to 12 weeks.
  Other Names: Wellbutrin XL, Forfivo XL, Zyban, and Aplenzin
  Arms: Group 5: Buproprion, Intense Counselling and NRT; Group 6: Buproprion, Intense Counselling; Group 7: Buproprion, Minimal Counselling and NRT; Group 8: Buproprion, Minimal Counselling
Drug: Long-acting nicotine replacement therapy — Nicotine replacement therapy (NRT) patches will be used daily from 1-10 weeks depending on participant's smoking history.
  Other Names: Transdermal nicotine
  Arms: Group 10: Nicotine, Intense Counselling; Group 11: Nicotine, Minimal Counselling and NRT; Group 12: Nicotine, Minimal Counselling; Group 9: Nicotine, Intense Counselling and NRT
Behavioral: Low-intensity counseling — A study coordinator or a member of the treatment team will provide a minimum level of initial counseling, approximately 10-20 minutes in length.
  Arms: Group 11: Nicotine, Minimal Counselling and NRT; Group 12: Nicotine, Minimal Counselling; Group 3: Varenicline, Minimal Counselling and NRT; Group 4: Varenicline, Minimal Counselling; Group 7: Buproprion, Minimal Counselling and NRT; Group 8: Buproprion, Minimal Counselling
Behavioral: High-intensity counseling — A counselor will provide eight sessions in the first 8 weeks of the study. Up to three follow up sessions over the next 4 months of study will be encouraged, but not required.
  Arms: Group 10: Nicotine, Intense Counselling; Group 1: Varenicline, Intense Counselling and NRT; Group 5: Buproprion, Intense Counselling and NRT; Group 6: Buproprion, Intense Counselling; Group 9: Nicotine, Intense Counselling and NRT; Group : Varenicline, Intense Counselling
Other: No nicotine replacement therapy — Participants in this group will not receive per required need nicotine replacement therapy.
  Other Names: nicotine gum, nicotine losenges, nicotine spray
  Arms: Group 10: Nicotine, Intense Counselling; Group 12: Nicotine, Minimal Counselling; Group 4: Varenicline, Minimal Counselling; Group 6: Buproprion, Intense Counselling; Group 8: Buproprion, Minimal Counselling; Group : Varenicline, Intense Counselling
Drug: Nicotine Replacement Products — Participants in this group will receive per required need nicotine replacement therapy.
  Other Names: nicotine gum, nicotine losenges, nicotine spray
  Arms: Group 11: Nicotine, Minimal Counselling and NRT; Group 1: Varenicline, Intense Counselling and NRT; Group 3: Varenicline, Minimal Counselling and NRT; Group 5: Buproprion, Intense Counselling and NRT; Group 7: Buproprion, Minimal Counselling and NRT; Group 9: Nicotine, Intense Counselling and NRT

SUMMARY:
Smoking cessation has been shown to improve the effectiveness and reduce the morbidity of tobacco-related cancer treatments. We will identify effective smoking cessation strategies for patients who are receiving treatment for tobacco-related cancer. In this trial, patients' preferences in smoking cessation therapy will be the principal determinant by providers in developing a three component regimen of pharmaceutical therapy, counseling, and nicotine replacement therapy. This study will identify this cohort's preferences for smoking cessation strategies. We will then examine the impact of utilizing patient preferences upon cessation efficacy by directly comparing cessation success in this study with our recently completed study of the same population using the same tobacco treatments which were randomly assigned.

DETAILED DESCRIPTION:
Background Cigarette smoking is associated with decreased survival and decreased efficacy of cancer therapy in those with smoking related malignancies. There is limited of study of smoking cessation for cancer patients being treated in regions with high tobacco use such as Kentucky. There is little study of cessation implementation in the community cancer treatment setting where the majority of cancer patients receive their cancer therapy. Most smokers have significant exposure to information and personal experience with tobacco treatments which, in some cases, leads to profound preferences. The effect of incorporating these patient preferences into tobacco treatment planning has not been studied or quantified.

Study Design Phase II therapeutic clinical trial.

Setting University of Kentucky Markey Cancer Center (MCC) and its affiliate research network of Community Cancer Centers (MCCRN)

Methods Ninety-three subjects will be selected. All subjects will be active smoking oncology patients with a diagnosis of smoking related malignancy who are beginning a new course of therapy. In conjunction with their treating clinician, all subjects will be counseled and then select one of 12 cessation strategies. This will include a choice of continuous pharmacologic agent (veranicline, bupropion or transdermal nicotine patch), counseling strategy (11 session high intensity motivational based counseling or single session low intensity counseling), and whether or not to use as needed nicotine (gum, lozenges or spray).

Data Analysis All subjects will be followed for six months. The primary endpoint will be a carbon monoxide monitoring confirmed negative seven-day point prevalence report of cessation at eight weeks. Data will then be analyzed and compared with a completed randomized clinical trial of the same treatment strategies in the same population of subjects where the cessation strategy was assigned (historical control). The proportion of subjects that have quit at week eight will be compared to the historical control proportion (namely, whether Ho:p=po vs Ha: p>po). This will be assessed using a z-score for a binomial proportion which will test whether the underlying proportion quitting at eight weeks (p) differs from the control proportion (po ranging from 0.215 to 0.26) estimated from our recently completed randomized trial of these same 12 cessation strategies.

Revised Enrollment Number: Effective with Amendment 2, Expand targeted enrollment from 96 to 126 due to higher than expected drop-out/censoring rate in order to evaluate the primary endpoint

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or recurrent tobacco related malignancy
* smoked at least 1 cigarette within 4 weeks of study enrollment
* 10-pack year history of cigarette smoking
* smoked at least 1 cigarette within 1 month of cancer diagnosis
* life expectancy greater than 1 year

Exclusion Criteria:

* allergy to buproprion, varenicline and transdermal medicine
* history of suicide attempt
* hospitalized for psychiatric illness within past 2 years
* history of active or uncontrolled eating disorder
* uncontrolled epilepsy or seizure disorder
* pregnant or lactating
* within 3 months of myocardial infarction
* unstable angina
* uncontrolled hypertension
* serious arrhythmia
* history of taking varenicline or buproprion within one month of enrollment
* concurrent enrollment in tobacco cessation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that quit smoking. | at week 8
  Proportion of participants that quit smoking at the 8 week assessment
Prevalence of cigarette use | at week 8
  Seven day point prevalence of cigarette use will be determined from participant reports and CO testing.

SECONDARY OUTCOMES:
Prevalence of cigarette use | 6 months
  Seven day point prevalence of cigarette use will be determined from participant reports and CO testing.
Preferred treatment | at baseline
  Proportion of participants preferring the treatment plan.
Change in Cigarette Use | 6 months
  Cigarette use will be recorded at weeks one, four, eight and at 6 months.
Drug Compliance | 6 months
  Subjects who complete 75% of the planned dosages of therapy will be considered compliant.
Counselling Compliance | 6 months
  Subjects who complete 60% of planned therapy sessions will be considered compliant.

OTHER OUTCOMES:
Number of patients requiring financial assistance with medication. | 6 months
  Number of patients requiring financial assistance with medication.
Number of patients with alteration in therapy | 6 months
  Number of patients with alteration in therapy due to ongoing cancer treatment.
Insurance coverage | 6 months
  Proportion of treatments covered by insurance/third party.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Valentino, MD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Med Center Health, Bowling Green, Kentucky
  - University Of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky

IPD SHARING:
Plan to Share IPD: No